CLINICAL TRIAL: NCT07342205
Title: A Prospective, Single-center, Randomized, Double-blind Controlled Study on the Treatment of Patients With Acute Lung Injury Caused by Sepsis Through Microbiota Transplantation
Brief Title: A Study on the Treatment of Patients With Acute Lung Injury Caused by Sepsis Through Microbiota Transplantation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Sun Yuting, Dr, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTEC-R-2025-44-1
Record Dates: First submitted 2025-08-31; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Acute Lung Injury(ALI); Sepsis Related Acute Lung Injury/Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Intervention Model Description: This study enrolled 60 patients with sepsis-related ALI who met the inclusion criteria. They were numbered using a random number table and randomly divided into Group A and Group B. Group A received basic treatment plus placebo (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, number: 250713-DZ), while Group B received basic treatment plus FMT (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, number: 250713-GT122. The donor screening followed international standards and there were no resistant bacteria or infectious pathogens). Note: Basic treatment included antibiotics, fluid resuscitation and respiratory support. Both groups received the corresponding bacterial solution and normal saline through the nasal intestinal tube, 100 mL each time, for 6 consecutive days. Oxygenation index (PaO2/FiO2), 28-day all-cause mortality rate and ICU hospitalization time were the main efficacy evaluation indicators. Adverse reactions ca
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of the clinical efficacy and mechanism of action of fecal microbiota transplantation (FMT (Placebo Comparator): The participants in this study will be divided into Group A and Group B. The participants in Group A will receive basic treatment and a placebo (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, serial number: 250713-DZ) for treatment.
  Interventions: Other: Placebo control group
- Human-derived active intestinal bacterial liquid (Experimental): The participants in Group B will receive basic treatment and human-derived active intestinal flora liquid (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, serial number: 250713-GT122) for treatment. Two groups were infused with the corresponding bacterial solution and the placebo bacterial solution through the nasal tube.
  Interventions: Other: Human-derived active intestinal bacterial liquid group

INTERVENTIONS:
Other: Placebo control group — The participants in Group A will receive basic treatment and placebo (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, serial number: 250713-DZ) for treatment.
  Arms: Evaluation of the clinical efficacy and mechanism of action of fecal microbiota transplantation (FMT
Other: Human-derived active intestinal bacterial liquid group — The participants in Group B will receive basic treatment and human-derived active intestinal flora liquid (provided by Shanghai Baoteng Medical Laboratory, specification: 50 mL per bottle, serial number: 250713-GT122) for treatment.
  Arms: Human-derived active intestinal bacterial liquid

SUMMARY:
Sepsis is a systemic inflammatory response syndrome triggered by infection, and it is a common critical illness in clinical practice, often leading to multiple organ dysfunction. Among these, acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are among the most severe complications. The mortality rate of sepsis-related lung injury is extremely high, reaching 30% - 50%. The existing treatment methods are unable to effectively reduce the high mortality rate of sepsis-related lung injury, and there are no specific treatment measures targeting lung injury itself. Dysbiosis of the intestinal flora plays an important role in the occurrence and development of sepsis-related lung injury. Fecal microbiota transplantation (FMT), as an effective means of regulating the intestinal flora, has shown certain therapeutic potential in some clinical studies. However, current research on FMT for treating sepsis-related lung injury is still in its infancy, and its mechanism is not yet fully clear. The clinical efficacy and safety also lack high-quality evidence support. Therefore, conducting this project's research will provide theoretical basis for targeted microecological treatment of sepsis-related lung injury; establishing a new strategy of combined microbiota transplantation technology for treating patients with sepsis ALI, and providing new ideas and methods for clinical treatment.

DETAILED DESCRIPTION:
Although certain research progress has been made in the pathogenesis and treatment of sepsis-related lung injury, many unresolved issues still exist. The existing treatment methods are unable to effectively reduce the high mortality rate of sepsis-related lung injury, and there are no specific treatment measures targeting the lung injury itself. Dysbiosis of the intestinal flora plays an important role in the occurrence and development of sepsis-related lung injury, and FMT, as an effective means of regulating the intestinal flora, has shown certain therapeutic potential in animal experiments and some clinical studies. However, current research on FMT for treating sepsis-related lung injury is still in its infancy, and its mechanism is not yet fully clear, and there is a lack of high-quality evidence to support its clinical efficacy and safety. Therefore, conducting this project's research is of great necessity. Through this project's research, it is expected to analyze the microbial-metabolism-immune regulatory network in the gut-lung axis, providing theoretical basis for targeted microecological treatment of sepsis-related lung injury; establish a new strategy for treating sepsis ALI patients using combined microbiota transplantation technology, and provide new ideas and methods for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Clear or suspected infection + SOFA score ≥ 2 points, and PaO₂/FiO₂ ≤ 300 mmHg;
* Capable of taking in nutrients (able to eat independently or receive enteral nutrition);
* Voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

* Indications for exclusion from FMT (Fecal Microbiota Transplantation) include massive gastrointestinal bleeding, intestinal obstruction, organic intestinal disorders, and severe damage to intestinal mucosa;
* Individuals with severe immune deficiencies, such as those with AIDS, leukemia, and those using immunosuppressive drugs;
* Pregnant women and lactating women;
* Those who cannot undergo nasal-intestinal catheterization or other transplantation methods;
* Patients who cannot cooperate to complete the study; Other situations where the researchers determine that a patient is not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation | 0-28 days
  Oxygenation index (PaO2/FiO2),
Efficacy evaluation | 0-28day
  28-day all-cause mortality rate
Efficacy evaluation | 0-28day
  ICU hospitalization time

SECONDARY OUTCOMES:
Inflammatory markers | (Day0, 3, 7, 14)
  The inflammatory biomarkers to be assessed include serum levels of C-reactive protein (CRP, measured in mg/L via immunoturbidimetric assay),
Vital signs (Day0 - 14) | Day 0，3，7，14
  Vital signs to be monitored as safety and physiological outcome measures
Changes in intestinal flora | Day0, 7, 28
  Changes in gut microbiota will be assessed as a secondary outcome by performing 16S ribosomal RNA gene sequencing on stool samples collected at baseline (pre-treatment),
Incidence of multi-drug resistant bacteria | Day0, 7, 28
  The primary/secondary outcome measure is the incidence of multidrug-resistant organism (MDRO) infection, defined as the proportion of patients who develop a new infection with bacteria resistant to at least one agent in three or more antimicrobial categories, confirmed by standard microbiological culture and antibiotic susceptibility testing.
Oxidative stress indicators | Day0, 3, 7, 14
  Oxidative stress biomarkers to be measured.
Functions of major organs | Day0, 3, 7, 14
  Myocardial enzyme profile outcome measures.
SOFA score | Day0, 3, 7, 14
  SOFA Score Calculation
Inflammatory markers | (Day0, 3, 7, 14)
  procalcitonin (PCT, measured in ng/mL via chemiluminescent immunoassay),
Inflammatory markers | (Day0, 3, 7, 14)
  tumor necrosis factor-alpha (TNF-α, measured in pg/mL via enzyme-linked immunosorbent assay).

CONTACTS AND LOCATIONS:
Locations (1):
- Putuo Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Putuo, China